CLINICAL TRIAL: NCT04447274
Title: A Single-arm, Open, Prospective, Single-center, Phase Ⅱ Clinical Study of Carilizumab Combined With Apatinib in theTtreatment of Advanced Inoperable Resection of Undifferentiated Pleomorphic Sarcoma and Alveolar Soft Tissue Sarcoma
Brief Title: A Study of Carilizumab in Combination With Apatinib in Subjects With Unresectable UPS and ASPS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, yihebali chi, Assistant Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPS and ASPS-IIT-SHR1210
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Sarcoma
Keywords: Camrelizumab; Apatinib; UPS; ASPS
MeSH Terms: conditions — Sarcoma | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab and Apatinib (Experimental): Drugs should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Camrelizumab and Apatinib

INTERVENTIONS:
Drug: Camrelizumab and Apatinib — Subject will receive SHR-1210 200mg every 2 weeks, with intravenous drip Apatinib 425 mg, oral, 5 consecutive days, 2 days off,each 14 day of a cycles

SUMMARY:
This study is a Single-arm, Open, Prospective, Single-center, Phase Ⅱ Clinical Study ,Target population is Advanced Inoperable Resection of Undifferentiated Pleomorphic Sarcoma (UPS) and Alveolar Soft Tissue Sarcoma (ASPS) .

The purpose of this study was to evaluate the safety and efficacy of combination of Camrelizumab and Apatinib in the treatment of unresectable UPS and ASPS

DETAILED DESCRIPTION:
In this study, eligible subject to accept study treatment. Camrelizumab combined with apatinib is a treatment cycle every 2 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Subjects >/= 16 years of age at the time of Informed Consent,male or female;
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
3. Life expectancy of at least three months;
4. Advanced undifferentiated pleomorphic sarcoma (UPS) confirmed by histopathology, patients who have failed in the first-line treatment and have progressed for 6 months; advanced acinar soft tissue sarcoma (ASPS) confirmed by histopathology, patients who have not been treated or who have failed in the first-line anti vascular drug treatment and progressed within 6 months;
5. Subjects enrolled must have measurable lesion(s) according to the RECIST 1.1 standard (the CT scan length of the tumor lesion > 10 mm;
6. All acute toxic reactions caused by previous anti-tumor treatment were relieved to 0-1 level before enrollment (according to NCI CTCAE 5.03) Version) or to the level specified in the inclusion / exclusion criteria (except for the toxicity that researchers think does not pose a safety risk to subjects, such as hair loss); if subjects undergo major surgery, they must have fully recovered from complications before starting treatment;
7. The main organ function is normal. All baseline laboratory requirements will be assessed and should be obtained within -14 days of randomization. Screening laboratory values must meet the following criteria.

   1. Hemoglobin ≥ 8.0 g/dL (90 g/L)
   2. Absolute neutrophil count ≥ 1.5× 109/L
   3. Platelets ≥ 80× 109/L
   4. Total bilirubin (TBIL) < 1.5 × upper limit of normal (ULN)
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × upper limit of normal(ULN);but < 5uln in patients with liver metastasis, alkaline phosphatase < 5 × ULN
   6. Serum creatinine ≤ 1× ULN or creatinine clearance > 45 mL/minute (using Cockcroft/Gault formula);
8. Women of childbearing age must have taken reliable contraceptive measures or carried out pregnancy test (serum or urine) within 7 days before entering the group, and the result is negative, and they are willing to use appropriate contraceptive methods during the test and 60 days after the last administration of test drugs. For men, they must agree to use appropriate methods of contraception or have undergone surgical sterilization during the trial period and within 120 days after the last administration of the trial drug;
9. Subjects should be voluntarily participate in clinical studies and informed consent should be signed.

Exclusion Criteria:

1. Known active central nervous system (CNS) metastasis and / or cancerous meningitis. Subjects who had previously received brain metastases may participate as long as they are stable and meet the following criteria: there is no evidence of imaging progress for at least four weeks prior to the first dose of trial treatment, and any neurological symptoms have returned to baseline, there is no evidence of new or expanded brain metastases, and steroids are not used for at least seven days prior to the trial treatment. This exception does not include cancerous meningitis, regardless of its clinical stability;
2. Immunosuppressive drugs were used within 14 days before the first use of carrizumab, excluding nasal spray and inhaled corticosteroids or systemic steroids with physiological dose (i.e. no more than 10 mg / day of prednisolone or other corticosteroids with physiological dose of the same drug); 3. Previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs for another stimulation or synergistic inhibition of T cell receptor (for example, CTLA-4, OX-40, CD137); 4. Uncontrollable hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg, despite systematic medication); 5. Severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poor control of arrhythmia (including QTc interval ≥ 450 ms for men and 470 MS for women); cardiac insufficiency of grade III-IV (according to NYHA classification of New York Heart Association, see Annex 3), or left ventricular ejection fraction (LVEF) < 50% indicated by color Doppler echocardiography; 6. Patients with any active autoimmune disease or history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism) shall not be included; 7. The subjects received systematic treatment such as bronchodilator, and the asthma control was not satisfactory and could not be included (the asthma in childhood has been completely relieved, and the adult can be included without any intervention); 8. Routine urine test indicated that urine protein was ≥ 1.0g, or 24-hour urine protein was ≥ 1.0g; 9. Abnormal coagulation (INR > 1.5 ULN or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolysis or anticoagulation treatment; Note: on the premise that the international standard ratio of prothrombin time (INR) is less than or equal to 1.5, it is allowed to use low-dose heparin (6000-12000 u daily for adults) or aspirin (less than or equal to 100 mg daily) for prevention purposes; 10. Severe infection (such as intravenous drip of antibiotics, antifungal drugs or antiviral drugs) occurred within 4 weeks before the first administration, or fever of unknown cause occurred during screening / before the first administration > 38.5 ° C; 11. Serious arteriovenous thrombotic events occurred in the first 12 months, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism; 12. In the first 4 weeks of the group, they had undergone major surgery or had severe traumatic injury, fracture or ulcer; 13. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active tuberculosis, active hepatitis B (HBV DNA ≥ 500 IU / ml), hepatitis C (HCV antibody positive, and HCV-RNA higher than the detection limit of the analysis method) or co infection with hepatitis B and C; 14. Patients with a clear history of allergy may be potentially allergic or intolerant to the biological agents of apatinib and carrizumab; 15. There are obvious factors affecting the absorption of oral drugs, such as inability to swallow, chronic diarrhea and intestinal obstruction. Or there were cavity organ sinus or perforation within 6 months; 16. Those who have a history of abuse of psychotropic substances and are unable to give up or have mental disorders; 17. Increase the risk associated with participating in the study or study drug, and other circumstances that, in the judgment of the investigator, may result in the patient not being eligible for inclusion in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free rate at 12 weeks (PFR 12weeks) | 12 weeks
  The RECIST 1.1 standard was used to evaluate the disease progression and the 12 week progression free rate was calculated.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | 6.5 months
  It is defined as the proportion of patients whose tumors shrink to a predetermined size and maintain a minimum time limit. It includes the cases of CR and PR
Progression free survival(PFS) | 6.5 months
  Refers to the date from the beginning of treatment to the first occurrence of disease progression or death caused by any reason, whichever occurs first
Duration of Response（DOR) | 6.5 months
  Time from the first assessment of Cr or PR to the first assessment of PD or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yihebali Chi, doctor, Principal Investigator — Chinese Academy of Medical Sciences